CLINICAL TRIAL: NCT06014801
Title: Low-Intensity Versus Medium-Intensity Continuous Kidney Replacement Therapy for Critically Ill Patients (LIMIT): a Multicenter Randomized Clinical Trial
Brief Title: Low-intensity Versus Medium-intensity Continuous Kidney Replacement Therapy for Critically Ill Patients
Acronym: LIMIT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jikei University School of Medicine (Other)
Collaborators: University of Fukui (Other); Tsuchiura Kyodo General Hospital (Other); Keio University (Other); Wakayama Medical University (Other); Jichi Medical University (Other); Sendai Medical Center (Unknown); Osaka Medical and Pharmaceutical University Hospital (Unknown)
Responsible Party: Principal Investigator, Tomoko Fujii, Professor, Jikei University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JKI23-002; jRCTs031230292 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury Requiring Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low intensity (Experimental): 12 mL/kg/hr
  Interventions: Drug: Dialysate fluid, Filtration replacement fluid
- Medium intensity (Active Comparator): 25 mL/kg/hr
  Interventions: Drug: Dialysate fluid, Filtration replacement fluid

INTERVENTIONS:
Drug: Dialysate fluid, Filtration replacement fluid — Dose of continuous hemodialysis and/or hemofiltration

SUMMARY:
This clinical trial aims to investigate whether the low treatment intensity (12 mL/kg/hr, low-dose hemodialysis/filtration) or the medium treatment intensity (25 mL/kg/hr, standard-dose hemodialysis/filtration) is more effective and safer for continuous renal replacement therapy in critically ill patients.

ELIGIBILITY:
Inclusion Criteria: Patient who meets all of the following criteria and who has given informed consent.

1. Adults (18 years of age or older, regardless of the time since ICU admission) currently admitted to an intensive care unit*.

   *Includes high care units, where continuous monitoring is conducted and intensive care physicians are in charge of medical care.
2. A diagnosis of acute kidney injury is made according to the Kidney Disease: Improving Global Outcomes (KDIGO) international diagnostic criteria (one of the following is met)

   * Serum creatinine increased by more than 0.3 mg/dL within 48 hours
   * Serum creatinine increased more than 1.5-fold from baseline and the increase is considered to have occurred within 7 days
   * Oliguria (< 0.5 mL/kg/hr) lasting more than 6 hours
3. The treating intensivist believes that continuous kidney replacement therapy is necessary

Exclusion Criteria: Patient who meets any of the following exclusion criteria will be excluded.

1. Receiving chronic dialysis or scheduled for initiation of chronic dialysis
2. Undergoing any kidney replacement therapy or blood purification therapy within 48 hours
3. When kidney replacement therapy using other dialysate or replacement fluids, such as citrate dialysis, is preferred due to coexisting bleeding disorders or allergy to acetate
4. Concomitant blood purification therapy other than hemofiltration/dialysis, such as plasma exchange
5. The patient is in a very critical condition and the treating physician believes that survival for more than 24 hours is unlikely
6. Previous participation in the study
7. After receiving a full explanation of the study and with full understanding, a patient do not consent to participate in the study of their own (or their substitute decision maker's) will.
8. The principal investigator (or an investigator) thinks it to be inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Composite of death and duration of kidney replacement therapy at 28 days | 28 days or hospital discharge whichever comes first
  Composite endpoint of death and duration of kidney replacement therapy at 28 days

SECONDARY OUTCOMES:
ICU mortality | 90 days or hospital discharge whichever comes first
Hospital mortality | 90 days or hospital discharge whichever comes first
Dialysis dependence at hospital discharge | 90 days or hospital discharge whichever comes first
28-day vasopressor-free days | 28 days or hospital discharge whichever comes first
28-day ventilator-free days | 28 days or hospital discharge whichever comes first
Serum creatinine level at the end of kidney replacement therapy | 90 days or hospital discharge whichever comes first
  Serum creatinine level on the day of final kidney replacement therapy and the day before
24-hour urine output at the end of kidney replacement therapy | 90 days or hospital discharge whichever comes first
  24-hour urine output on the day of final kidney replacement therapy and the day before

OTHER OUTCOMES:
Hypokalemia | up to 7 days of continuous kidney replacement therapy
Hypophosphatemia | up to 7 days of continuous kidney replacement therapy
Sodium bicarbonate solutions that administered | up to 7 days of continuous kidney replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Fujii, MD,PhD, Study Chair — Jikei University School of Medicine
Locations (9):
- Japan (9):
  - Sendai Medical Center, Sendai, Miyagi
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - University of Fukui Hospital, Fukui
  - Tsuchiura Kyodo General Hospital, Ibaraki
  - Osaka University Hospital, Osaka
  - Jichi Medical University Hospital, Tochigi
  - Jikei University Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Beaubien-Souligny W, Thompson Bastin M, Teixeira JP, Cerda J, Connor MJ Jr, Dijanic Zeidman A, Garimella PS, Juncos L, Lopez-Ruiz A, Mehta R, Reis T, Rizo-Topete L, Silver SA, Da Silva JR, Speer R, Vijayan A, Wells C, Wille K, Yessayan L, Tolwani A, Neyra JA. Proceedings of the University of Alabama at Birmingham Continuous Renal Replacement Therapy Academy (2023-2024): Managing De-Escalation of Acute Renal Replacement Therapy and Optimizing Drug Dosing during Renal Replacement Therapy Transitions. Kidney360. 2025 Oct 1;6(10):1798-1809. doi: 10.34067/KID.0000000951. Epub 2025 Aug 8. PMID 40779331